CLINICAL TRIAL: NCT07031687
Title: Effects and Mechanisms of Temporal Interference Brain Stimulation on Memory Function in Preclinical Alzheimer's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Ying Han, Professor, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TIBS_hanying_0605
Record Dates: First submitted 2025-06-06; First posted 2025-06-22 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalized Closed-Loop Temporal Interference Brain Stimulation (Experimental): Participants in this arm will receive active TIBS targeted at the bilateral hippocampus. Stimulation parameters include a 5 Hz (Theta band) low-frequency modulation envelope, generated by two high-frequency current pairs (e.g., f1=2000 Hz, f2=2005 Hz). Peak-to-peak current intensity for each pair will be 2 mA (or 1 mA per electrode). Stimulation will be delivered daily for 40 minutes, 6 days/week, for a total of 2 weeks. Individualized targeting and initial intensity optimization will be guided by baseline sMRI and DTI. Real-time high-density EEG monitoring during each daily session (D2-D11) will provide feedback on brain activity (e.g., EEG power spectra, functional connectivity features) to enable closed-loop optimization of transcranial stimulation intensity and phase parameters.
  Interventions: Device: Active TIBS
- Sham Temporal Interference Brain Stimulation (Sham Comparator): Participants in this arm will receive sham stimulation designed to mimic the sensation of active TIBS without therapeutic output. This will involve using a sham coil or a device mode with extremely low current intensity (e.g., 0.1-0.2 mA) or brief ramp-up/ramp-down sensations at the beginning and end of sessions, with no effective current delivery during the main stimulation period. The stimulation position and apparent parameters will be identical to the active TIBS group to maintain blinding.
  Interventions: Device: Sham TIBS

INTERVENTIONS:
Device: Active TIBS — Participants receive active TIBS targeted at the bilateral hippocampus. Stimulation parameters include a 5 Hz (Theta band) low-frequency modulation envelope, generated by two high-frequency current pairs (e.g., f1=2000 Hz, f2=2005 Hz). Peak-to-peak current intensity for each pair will be 2 mA (or 1 mA per electrode). Stimulation is delivered daily for 40 minutes, 6 days/week, for a total of 2 weeks. Individualized targeting and initial intensity optimization are guided by baseline sMRI and DTI. Real-time high-density EEG monitoring during each daily session (D2-D11) provides feedback on brain activity
  Arms: Personalized Closed-Loop Temporal Interference Brain Stimulation
Device: Sham TIBS — Participants receive sham stimulation designed to mimic the sensation of active TIBS without therapeutic output. This involves using a sham coil or a device mode with extremely low current intensity (e.g., 0.1-0.2 mA) or brief ramp-up/ramp-down sensations at the beginning and end of sessions, with no effective current delivery during the main stimulation period. The stimulation position and apparent parameters are identical to the active TIBS group to maintain blinding.
  Arms: Sham Temporal Interference Brain Stimulation

SUMMARY:
The goal of this clinical trial is to learn if personalized, multimodal imaging-guided, EEG-based closed-loop Temporal Interference Brain Stimulation (TIBS) can improve memory function in individuals with preclinical Alzheimer's Disease (AD).

The main questions it aims to answer are:

1. Does personalized TIBS lead to significant changes in functional connectivity strength of hippocampal-cortical networks at the end of the 2-week intervention compared to baseline?
2. What are the short-term (end of 2-week intervention) and medium-to-long-term (4 weeks and 12 weeks post-intervention) effects of personalized TIBS on episodic and working memory, as well as other cognitive domains in preclinical AD?
3. How does personalized TIBS modulate brain activity and connectivity, as measured by EEG power spectra and functional MRI (fMRI) functional connectivity, in preclinical AD?
4. What is the safety profile of personalized TIBS in this population?

Researchers will compare participants receiving active personalized TIBS to participants receiving sham (inactive) stimulation to see if TIBS effectively improves memory function and induces neural plasticity.

Participants will:

1. Undergo initial screening including neuropsychological assessments and blood p-tau217 testing to identify preclinical AD.
2. Receive either active personalized TIBS or sham stimulation daily for 40 minutes, 6 days a week, for 2 weeks.
3. Have individualized TIBS parameters (e.g., target localization, intensity) determined using baseline structural MRI and DTI.
4. Undergo real-time high-density EEG monitoring during daily stimulation sessions to enable closed-loop adjustment of stimulation parameters.
5. Participate in follow-up assessments at the end of the 2-week intervention, and at 4 weeks and 12 weeks post-intervention.
6. Receive multimodal imaging (sMRI, rs-fMRI, task-fMRI, DTI) and blood biomarker assessments at various time points.
7. Receive Aβ-PET and tau-PET scans, along with comprehensive neuropsychological assessments, at the 12-week follow-up.
8. Have their safety continuously monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals recruited from neurology memory clinics or communities.
* Age between 60 and 80 years old, inclusive; no gender limitation.
* Right-handed.
* Cognitive function test results within normal range after age, gender, and education-level adjustment, OR mild cognitive impairment not yet meeting diagnostic criteria for Mild Cognitive Impairment (MCI), OR only subjective cognitive decline.
* Individuals classified as preclinical AD based on the revised 2024 AD diagnostic and staging criteria (i.e., cognitively normal with positive plasma p-tau217 or positive Aβ PET).
* Full understanding of the study, voluntary participation, and provision of written informed consent approved by the Ethics Committee.

Exclusion Criteria:

* Past or present neurological diseases (e.g., stroke, epilepsy, Parkinson's disease, multiple sclerosis).
* Psychiatric disorders such as severe depression or severe anxiety.
* Systemic diseases causing cognitive decline (e.g., severe thyroid dysfunction, severe liver or kidney disease, severe nutritional deficiencies).
* Currently taking medications that may affect cognitive function (e.g., anticholinergics, benzodiazepines, antipsychotics) that cannot be discontinued or adjusted.
* Other factors leading to cognitive decline that are not AD-related.
* Contraindications for MRI scans, such as claustrophobia, implanted metallic devices (e.g., pacemakers, cochlear implants, aneurysm clips), or history of head injury with retained metal fragments.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Functional Connectivity Strength of Hippocampal-Cortical Networks | Baseline, End of 2-week intervention.
  Quantified by resting-state fMRI (rs-fMRI) functional connectivity strength within and between key memory-related networks (e.g., default mode network, hippocampal-cortical network) at the end of the 2-week intervention. Specific metrics will include ALFF, ReHo, FCS, and ACF.

SECONDARY OUTCOMES:
Changes from Baseline in Hippocampal Gray Matter Density (sMRI) | Baseline, End of 2-week intervention, 4 weeks post-intervention, 12 weeks post-intervention
  Evaluation of changes in hippocampal gray matter density or volume, quantified using structural Magnetic Resonance Imaging (sMRI). This measure assesses the structural integrity and potential atrophy or increase in gray matter in a key brain region associated with memory.
Changes from Baseline in Cortical Thickness (sMRI) | Baseline, End of 2-week intervention, 4 weeks post-intervention, 12 weeks post-intervention
  Evaluation of changes in cortical thickness across various brain regions, quantified using structural Magnetic Resonance Imaging (sMRI). This measure assesses the integrity and potential thinning or thickening of the cerebral cortex.
Changes from Baseline in Resting-State Functional Connectivity (fMRI) | Baseline, 4 weeks post-intervention, 12 weeks post-intervention
  Evaluation of changes in resting-state functional connectivity using functional Magnetic Resonance Imaging (fMRI). This assesses the temporal correlations between spontaneous fluctuations in BOLD signals across different brain regions, reflecting synchronized neural activity. Specific brain networks (e.g., Default Mode Network, Salience Network) or seed-based connectivity will be analyzed.
Changes from Baseline in White Matter Integrity (DTI) | Baseline, End of 2-week intervention, 4 weeks post-intervention, 12 weeks post-intervention
  Evaluation of changes in white matter integrity, assessed using Diffusion Tensor Imaging (DTI). Key metrics to be analyzed include Fractional Anisotropy (FA), Mean Diffusivity (MD), Axial Diffusivity (AD), and Radial Diffusivity (RD), reflecting the directionality and magnitude of water diffusion in white matter tracts.
Changes from Baseline in AD Molecular Pathologies and Blood Biomarkers | Baseline, 12 weeks post-intervention
  Evaluation of brain amyloid-beta (Aβ) deposition via Aβ-PET imaging, brain tau pathology via tau-PET imaging, and dynamic changes in plasma biomarkers (e.g., p-tau217, Aβ42/40 ratio, NfL, GFAP, α-synuclein, BDNF).
Changes from Baseline in Auditory Verbal Learning Test-H (AVLT-H) Score | Baseline, End of 2-week intervention, 4 weeks post-intervention, 12 weeks post-intervention
  Measures episodic memory. The Auditory Verbal Learning Test - Delayed Recall (AVLT-H) score typically represents the number of words recalled after a delay.
  Full Scale Name: Auditory Verbal Learning Test-H Minimum Value: 0 Maximum Value: Delayed Recall--12; Recognition--24 Higher Scores Mean: Better memory.
Changes from Baseline in n-back Task Performance Score | Baseline, End of 2-week intervention, 4 weeks post-intervention, 12 weeks post-intervention
  Measures working memory. Performance on the n-back task is typically measured by accuracy (percentage of correct responses) or the highest 'n' level achieved.
  Full Scale Name: n-back Task Performance Minimum Value: 0% accuracy or lowest 'n' level Maximum Value: 100% accuracy or highest 'n' level tested Higher Scores Mean: Better working memory.
Changes from Baseline in Mini-Mental State Examination (MMSE) Score | Baseline, End of 2-week intervention, 4 weeks post-intervention, 12 weeks post-intervention
  Measures global cognitive function. Full Scale Name: Mini-Mental State Examination (MMSE) Minimum Value: 0 Maximum Value: 30 Higher Scores Mean: A better global cognitive function.
Changes from Baseline in Montreal Cognitive Assessment - Basic (MoCA-B) Score | Baseline, End of 2-week intervention, 4 weeks post-intervention, 12 weeks post-intervention
  Measures global cognitive function. Full Scale Name: Montreal Cognitive Assessment - Basic (MoCA-B) Minimum Value: 0 Maximum Value: 30 Higher Scores Mean: A better global cognitive function.
Changes from Baseline in Verbal Fluency Test Score | Baseline, End of 2-week intervention, 4 weeks post-intervention, 12 weeks post-intervention
  Measures language function. The score represents the number of words generated. Full Scale Name: Verbal Fluency Test Minimum Value: 0 Maximum Value: None Higher Scores Mean: A better verbal fluency.
Changes from Baseline in Boston Naming Test (BNT) Score | Baseline, End of 2-week intervention, 4 weeks post-intervention, 12 weeks post-intervention
  Measures language function. The score represents the number of words generated. Full Scale Name: Boston Naming Test Minimum Value: 0 Maximum Value: 30 Higher Scores Mean: A better naming ability.
Changes from Baseline in Shape trails test A&B (STT-A&B) Score | Baseline, End of 2-week intervention, 4 weeks post-intervention, 12 weeks post-intervention
  Measures visual scanning and motor speed. The score is the time taken to complete the task.
  Full Scale Name: Shape trails test Minimum Value: 0 Maximum Value: None Higher Scores Mean: Slower completion time
Incidence and Severity of Adverse Events (AEs) | through study completion, an average of 14 weeks
  Monitoring and reporting of all adverse events and serious adverse events related to the intervention, including their frequency, severity, and relationship to the study intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ying Han, PhD, Principal Investigator — Xuanwu Hospital of Capital Medical University
Locations (2):
- China (2):
  - Hainan university, Sanya, Hainan
  - Xuanwu Hospital of Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lv X, Cheng Z, Wang Q, Gao F, Dai L, Du C, Liu C, Xie Q, Shen Y, Shi J; China Aging and Neurodegenerative Initiative (CANDI) Consortium. High burdens of phosphorylated tau protein and distinct precuneus atrophy in sporadic early-onset Alzheimer's disease. Sci Bull (Beijing). 2023 Nov 30;68(22):2817-2826. doi: 10.1016/j.scib.2023.10.019. Epub 2023 Oct 27. PMID 37919158
- [Background] Chen Q, Chen F, Long C, Zhu Y, Jiang Y, Zhu Z, Lu J, Zhang X, Nedelska Z, Hort J, Zhang B. Spatial navigation is associated with subcortical alterations and progression risk in subjective cognitive decline. Alzheimers Res Ther. 2023 Apr 25;15(1):86. doi: 10.1186/s13195-023-01233-6. PMID 37098612
- [Background] Zhao K, Wang D, Wang D, Chen P, Wei Y, Tu L, Chen Y, Tang Y, Yao H, Zhou B, Lu J, Wang P, Liao Z, Chen Y, Han Y, Zhang X, Liu Y. Macroscale connectome topographical structure reveals the biomechanisms of brain dysfunction in Alzheimer's disease. Sci Adv. 2024 Oct 11;10(41):eado8837. doi: 10.1126/sciadv.ado8837. Epub 2024 Oct 11. PMID 39392880
- [Background] Violante IR, Alania K, Cassara AM, Neufeld E, Acerbo E, Carron R, Williamson A, Kurtin DL, Rhodes E, Hampshire A, Kuster N, Boyden ES, Pascual-Leone A, Grossman N. Non-invasive temporal interference electrical stimulation of the human hippocampus. Nat Neurosci. 2023 Nov;26(11):1994-2004. doi: 10.1038/s41593-023-01456-8. Epub 2023 Oct 19. Erratum In: Nat Neurosci. 2023 Dec;26(12):2252. doi: 10.1038/s41593-023-01517-y. PMID 37857775
- [Background] Vassiliadis P, Beanato E, Popa T, Windel F, Morishita T, Neufeld E, Duque J, Derosiere G, Wessel MJ, Hummel FC. Non-invasive stimulation of the human striatum disrupts reinforcement learning of motor skills. Nat Hum Behav. 2024 Aug;8(8):1581-1598. doi: 10.1038/s41562-024-01901-z. Epub 2024 May 29. PMID 38811696
- [Background] Beanato E, Moon HJ, Windel F, Vassiliadis P, Wessel MJ, Popa T, Pauline M, Neufeld E, De Falco E, Gauthier B, Steiner M, Blanke O, Hummel FC. Noninvasive modulation of the hippocampal-entorhinal complex during spatial navigation in humans. Sci Adv. 2024 Nov;10(44):eado4103. doi: 10.1126/sciadv.ado4103. Epub 2024 Oct 30. PMID 39475597
- [Background] Grossman N, Bono D, Dedic N, Kodandaramaiah SB, Rudenko A, Suk HJ, Cassara AM, Neufeld E, Kuster N, Tsai LH, Pascual-Leone A, Boyden ES. Noninvasive Deep Brain Stimulation via Temporally Interfering Electric Fields. Cell. 2017 Jun 1;169(6):1029-1041.e16. doi: 10.1016/j.cell.2017.05.024. PMID 28575667
- [Background] Jack CR Jr, Andrews JS, Beach TG, Buracchio T, Dunn B, Graf A, Hansson O, Ho C, Jagust W, McDade E, Molinuevo JL, Okonkwo OC, Pani L, Rafii MS, Scheltens P, Siemers E, Snyder HM, Sperling R, Teunissen CE, Carrillo MC. Revised criteria for diagnosis and staging of Alzheimer's disease: Alzheimer's Association Workgroup. Alzheimers Dement. 2024 Aug;20(8):5143-5169. doi: 10.1002/alz.13859. Epub 2024 Jun 27. PMID 38934362